CLINICAL TRIAL: NCT07239934
Title: Diagnostic Role of Gastrointestinal Endoscopy in Assiut University Children Hospital
Brief Title: Pediatric GI Endoscopy at Assiut University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Shaban Mohamed Farghly, Resident of Pediatrics, Assiut University Children's Hospital, Assiut University
Other Study IDs: endoscopy in AUCH
Record Dates: First submitted 2025-09-23; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Diarrhea; Persistent Vomitting; Gastrointestinal Bleeding; Dysphagia; Foreign Body Ingestion; Failure to Thrive; Pediatric Inflammatory Bowel Disease
Keywords: pediatric gastrointestinal endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Deglutition Disorders; Failure to Thrive | interventions — Endoscopy, Gastrointestinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Gastrointestinal Endoscopy — Children undergoing evaluation for gastrointestinal symptoms (such as abdominal pain, bleeding, vomiting, chronic diarrhea, suspected foreign body ingestion, or growth failure) will undergo diagnostic gastrointestinal endoscopy (upper or lower as clinically indicated). The procedure will be performed under appropriate sedation/anesthesia using a standard pediatric endoscope. During endoscopy, visualization of the mucosa will be carried out, and biopsies may be taken if needed for histopathological examination.

SUMMARY:
1. To evaluate the diagnostic role, and outcomes of upper and lower gastrointestinal (GI) endoscopy in identifying gastrointestinal disorders among infants and pediatric patients attending Assiut University Children Hospital.
2. To determine which pediatric patients require endoscopy as part of the diagnostic process.
3. To assess the safety and effectiveness of endoscopic procedures in the detection and management of various gastrointestinal disorders among pediatric patients at Assiut University Children Hospital.

DETAILED DESCRIPTION:
Pediatric endoscopy plays a pivotal role in the diagnosis and management of various gastrointestinal and hepatological disorders in children.It allows doctors to see inside the digestive system, identify problems, and sometimes even treat them during the same procedure. It is a rapidly evolving field, with continuous advancements in both endoscopic technology and procedural skills, making it a safe, effective, and reliable diagnostic and therapeutic tool. Today, pediatric endoscopy is considered an essential part of evaluating and treating a wide range of gastrointestinal conditions in children. Accurate and timely diagnosis of gastrointestinal disorders is critical to prevent complications, reduce morbidity, and ensure appropriate management. These disorders are among the most common health problems affecting children worldwide. They often present with a wide variety of symptoms, including failure to thrive, unexplained anemia, recurrent vomiting, dysphagia (difficulty swallowing), acute epigastric pain, foreign body ingestion, hematemesis (vomiting blood), melena (black, tarry stools), abdominal pain, rectal bleeding, bloody diarrhea, and chronic diarrhea. At Assiut University Children Hospital, a major tertiary care center serving Upper Egypt. In recent years, there has been growing use of gastrointestinal endoscopy as a main method for diagnosing and treating various GI conditions. IT includes foreign body removal, management of caustic ingestion injuries, treatment of esophageal strictures, assessment of gastroesophageal reflux disease (GERD) severity, diagnosis of Helicobacter pylori infection through endoscopic biopsy, evaluation of eosinophilic esophagitis, management of variceal and non-variceal gastrointestinal bleeding such as deep ulcerations and gastroduodenal vascular malformations. In addition, ileocolonoscopy is commonly performed to assess lower gastrointestinal disorders such as juvenile polyps, inflammatory bowel disease (IBD), allergic colitis, vascular malformations, and infectious colitis.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 1day to 18 years undergoing diagnostic endoscopy.

Exclusion Criteria:

* Incomplete patient data.
* Patients undergoing follow-up procedures.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to Assiut University Children Hospital who present with gastrointestinal symptoms (such as abdominal pain, vomiting, hematemesis, melena, diarrhea, or unexplained anemia) and are referred for diagnostic gastrointestinal endoscopy as part of their clinical evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of gastrointestinal endoscopy | Within 30 days after endoscopy.
  Proportion (%) of pediatric patients in whom gastrointestinal endoscopy provides a definitive diagnosis based on endoscopic and histopathological findings.
Distribution of clinical indications for pediatric endoscopy | At the time of endoscopy.
  Proportion (%) of children undergoing endoscopy for each indication (e.g., abdominal pain, GI bleeding, chronic diarrhea).
Correlation between clinical suspicion and confirmed diagnosis | Within 30 days after endoscopy.
  Level of agreement between pre-procedure clinical suspicion and final diagnosis based on endoscopic and histopathological findings (reported as percentage concordance).

SECONDARY OUTCOMES:
Types and frequencies of gastrointestinal disorders diagnosed by endoscopy | Within 30 days after endoscopy.
  Frequency distribution of gastrointestinal disorders diagnosed in pediatric patients undergoing endoscopy.
Safety and complication rates of pediatric endoscopy | From the time of endoscopy until 7 days post-procedure.
  Incidence (%) of procedure-related complications (e.g., bleeding, perforation, infection).
change in awareness among healthcare providers | Up to 6 months from start of study.
  Change in awareness and knowledge about pediatric gastrointestinal endoscopy, assessed by structured questionnaire score before and after educational sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abd elaziz, MD, Study Director — Assiut University, Faculty of Medicine, Children Hospital; rehab ibrahim, MD, Study Director — Assiut University, Faculty of Medicine, Children Hospital
Locations (1):
- Endoscopic Centre at Assiut University Children Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bohara TP, Laudari U, Thapa A, Rupakheti S, Joshi MR. Appropriateness of Indications of Upper Gastrointestinal Endoscopy and its Association With Positive Finding. JNMA J Nepal Med Assoc. 2018 Jan-Feb;56(209):504-509. PMID 30058633
- [Result] Schluckebier D, Afzal NA, Thomson M. Therapeutic Upper Gastrointestinal Endoscopy in Pediatric Gastroenterology. Front Pediatr. 2022 Feb 25;9:715912. doi: 10.3389/fped.2021.715912. eCollection 2021. PMID 35280448
- [Result] Tringali A, Thomson M, Dumonceau JM, Tavares M, Tabbers MM, Furlano R, Spaander M, Hassan C, Tzvinikos C, Ijsselstijn H, Viala J, Dall'Oglio L, Benninga M, Orel R, Vandenplas Y, Keil R, Romano C, Brownstone E, Hlava S, Gerner P, Dolak W, Landi R, Huber WD, Everett S, Vecsei A, Aabakken L, Amil-Dias J, Zambelli A. Pediatric gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) and European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) Guideline Executive summary. Endoscopy. 2017 Jan;49(1):83-91. doi: 10.1055/s-0042-111002. Epub 2016 Sep 12. PMID 27617420
- [Result] Fachler T, Shteyer E, Orlanski Meyer E, Shemasna I, Lev Tzion R, Rachman Y, Bergwerk A, Turner D, Ledder O. Pediatric Gastrointestinal Endoscopy: Diagnostic Yield and Appropriateness of Referral Based on Clinical Presentation: A Pilot Study. Front Pediatr. 2021 Oct 29;9:607418. doi: 10.3389/fped.2021.607418. eCollection 2021. PMID 34778118
- [Result] Ngo PD, Lightdale JR. Advances in Pediatric Endoscopy. Gastroenterol Clin North Am. 2024 Dec;53(4):539-555. doi: 10.1016/j.gtc.2024.08.010. Epub 2024 Sep 30. PMID 39489574
- [Result] Franciosi JP, Fiorino K, Ruchelli E, Shults J, Spergel J, Liacouras CA, Leonard M. Changing indications for upper endoscopy in children during a 20-year period. J Pediatr Gastroenterol Nutr. 2010 Oct;51(4):443-7. doi: 10.1097/MPG.0b013e3181d67bee. PMID 20562722